CLINICAL TRIAL: NCT00788619
Title: Use of Nitric Oxide Metabolites for Predicting Embryo Quality in In-Vitro Fertilization
Brief Title: Use of Nitric Oxide Metabolites for Predicting Embryo Quality in In-Vitro Fertilization (IVF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty with recruitment
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00013752
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Infertility
Keywords: Infertility; Assisted reproductive technology; Nitric oxide
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 3 transfer (Active Comparator): Subjects in this arm will have two embryos transferred three days after fertilization. Embryos will be selected based on the concentration of nitric oxide metabolites in the culture medium.
  Interventions: Procedure: Transfer of embryos on day 3 or day 5 after fertilization.
- Day 5 transfer (Active Comparator): Subjects will have two embryos transferred on day 5 after fertilization with selection of embryos based on morphologic criteria.
  Interventions: Procedure: Day 5 transfer

INTERVENTIONS:
Procedure: Transfer of embryos on day 3 or day 5 after fertilization. — Subjects will be allocated at random to the two arms. Group 1 will have two embryos transferred on day 3 based on nitric oxide concentration. Group 2 will have two embryos transferred on day 5 based on morphologic criteria.
  Arms: Day 3 transfer
Procedure: Day 5 transfer — Subjects will have embryo transfer on day 5 after fertilization. Selection of embryos to transfer will be based on morphologic criteria.
  Arms: Day 5 transfer

SUMMARY:
Improvements in In-Vitro Fertilization (IVF) outcomes have largely been due to the generation of excess embryos allowing for multiple embryo transfer. Unfortunately this has also increased the risk of multiple pregnancy with associated maternal and neonatal morbidity and mortality. The investigators believe that the concentration of nitric oxide metabolites measured in the culture medium from the first day of culture can identify the best quality embryos allowing us to transfer a limited number of embryos without compromising the optimum chance for pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-37
* Female
* Less than two previous unsuccessful IVF cycles

Exclusion Criteria:

* Day 3 FSH >9.9
* Fewer than 8 mature oocytes retrieved
* Fewer than 8 normally fertilized embryos on day 2 after fertilization

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with viable pregnancy one month after embryo transfer | 1 month

SECONDARY OUTCOMES:
Percentage of subjects with > 2 viable embryos one month after embryo transfer | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Kolp, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Fertility Center, Lutherville, Maryland, United States